CLINICAL TRIAL: NCT06848920
Title: Phase II Clinical Study of Sinibolimab Combined with Lenvatinib As Neoadjuvant Therapy for Locally Advanced Unresectable Differentiated Thyroid Carcinoma
Brief Title: Study of Sinibolimab Combined with Lenvatinib As Neoadjuvant Therapy for Locally Advanced Unresectable Differentiated Thyroid Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiongfei Yu, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024102
Record Dates: First submitted 2025-01-26; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Differentiated Thyroid Carcinoma (DTC); Neoadjuvant Therapy
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Sinibolimab combined with Lenvatinib group
  Interventions: Drug: Immunotherapy combined with Multikinase inhibitors in neoadjuvant treatment

INTERVENTIONS:
Drug: Immunotherapy combined with Multikinase inhibitors in neoadjuvant treatment — Sinibolimab combined with Lenvatinib in neoadjuvant treatment

SUMMARY:
This study is a single-arm, prospective investigation aimed at evaluating the efficacy of Sinibolimab combined with Lenvatinib as neoadjuvant therapy for locally advanced unresectable differentiated thyroid carcinoma in a Phase II clinical trial. The study plans to enroll 20 patients with locally advanced unresectable papillary thyroid carcinoma. Eligible participants will receive a combination of Sinibolimab and Lenvatinib for four cycles. After completing the four cycles of treatment, the tumor response will be assessed to determine the feasibility of surgical intervention. Participants who complete treatment will enter a follow-up period for safety monitoring and survival assessment. The primary endpoints of the study include the major pathological response (MPR) and the R0/R1 resection rate. Secondary endpoints include the objective response rate (ORR) after four cycles, 1-year and 2-year disease-free survival (DFS) rates, serious adverse events (SAE), and immune-related adverse events (irAE).

DETAILED DESCRIPTION:
This study is a single-arm, prospective Phase II clinical trial designed to evaluate the efficacy and safety of Sinibolimab in combination with Lenvatinib as a neoadjuvant therapy for patients with locally advanced, unresectable differentiated thyroid carcinoma (DTC). A total of 20 patients with locally advanced unresectable papillary thyroid carcinoma (PTC) meeting eligibility criteria will be enrolled. Participants will receive four cycles of the combination therapy consisting of Sinibolimab, a PD-1 inhibitor, and Lenvatinib, a tyrosine kinase inhibitor known for its anti-angiogenic and anti-proliferative properties.

After completing the four treatment cycles, tumor response will be evaluated using imaging and pathological assessments to determine if surgical resection of the tumor becomes feasible. The primary endpoints are the major pathological response (MPR) after neoadjuvant therapy and the R0/R1 resection rate, which measures the proportion of patients achieving complete or near-complete tumor removal.

Secondary endpoints include objective response rate (ORR), defined as the proportion of patients exhibiting a measurable reduction in tumor size after four cycles, as well as 1-year and 2-year disease-free survival (DFS) rates. Additionally, the trial will comprehensively monitor treatment-related safety, focusing on the incidence of serious adverse events (SAEs) and immune-related adverse events (irAEs). Patients who complete the trial will enter a post-treatment follow-up phase to evaluate long-term outcomes, including survival and late-onset adverse effects.

This investigation will provide insight into the potential of Sinibolimab combined with Lenvatinib to convert unresectable tumors into resectable states, thereby improving therapeutic options for patients with advanced thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed or recurrent locally advanced (T4N1M0) differentiated thyroid carcinoma with an estimated risk of R2 resection.

Performance Status (PS) score of 0-1. Age ≥ 18 years. Measurable lesions according to RECIST 1.1 criteria. Normal function of major organ systems.

Exclusion Criteria:

* Intratracheal airway tumors. Complete carotid artery encasement/invasion. Full-thickness infiltration of the esophageal wall. Arterial thrombosis/cancer thrombus. Active hemoptysis (bright red blood ≥ 1/2 teaspoon) or other uncontrolled bleeding within 21 days prior to study enrollment.

History of prior neck radiotherapy. Previous treatment with Lenvatinib or immunotherapy. Participants with > 1+ proteinuria on urine dipstick will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥ 1g/24 hours will be ineligible.

Active, known, or suspected autoimmune diseases. Participants requiring long-term systemic corticosteroid therapy. Participants using bronchodilators, inhaled corticosteroids intermittently due to COPD or asthma, or those receiving local corticosteroid injections may be eligible.

Active unstable angina and/or congestive heart failure. New-onset myocardial infarction within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | After four cycles of treatment（each cycle is 21 days）
R0/R1 resection rate | After four cycles of treatment（each cycle is 21 days）
  R0 (no tumor at the surgical margins) / R1 (microscopically negative surgical margins) resection rates.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF